CLINICAL TRIAL: NCT01602991
Title: Sensitivity, Specificity, and Positive and Negative Predictive Values of Clinic-based Nasopharyngoesophagogastroscopy Following Bariatric Surgery
Brief Title: Clinic-based Nasopharyngoesophagogastroscopy Following Bariatric Surgery
Acronym: EGScan
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: difficulty obtaining funding
Sponsor: Dennis Hong MD (Other)
Collaborators: Vantage Endoscopy (Unknown)
Responsible Party: Sponsor-Investigator, Dennis Hong MD, PI, McMaster University
Organization: McMaster University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 12-3647
Record Dates: First submitted 2012-05-07; First posted 2012-05-21 (Estimated); Last update posted 2015-09-24 (Estimated); Status verified 2015-09

CONDITIONS: Obesity
Keywords: Obesity; Endoscopy; Nasopharyngoesophagogastroscopy; Bariatric Surgery; Gastric Bypass Surgery
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: clinic-based nasopharyngoendoscopy — The study intervention is an in-office transnasal esophagoscopy. It is done in clinic, immediately after deciding the patient requires investigation of their upper gastrointestinal tract and the patient signs consent. The nasopharynx and oral pharynx is topically anesthetized. Since flexible scope is much thinner than a standard endoscopy, there is no requirement for intravenous sedation and thus, no requirement for specialized monitoring, nursing or recovery units. The procedure takes approximately 10 minutes. This study will be using the E.G. Scan II System.
  Other Names: E.G. Scan
Procedure: Standard Endoscopy — The control procedure is standard endoscopy. Endoscopy will be performed as per standard clinic practice. It is typically scheduled within 2 weeks of seeing the patient in clinic. The patient will be required to fast for 6 hours prior to the procedure. In most cases, patients will require intravenous sedation. If sedation is used, the patient will be required to take the day off work and have someone drive them home. This is the standard treatment for patients who present with upper gastrointestinal symptoms post-bariatric surgery. Patients who choose not to participate in this study will still undergo endoscopy as per standard clinical practice.

SUMMARY:
This study aims to determine that this new technology, nasopharyngoendoscopy, is just as effective in diagnosing problems as the current gold standard.

DETAILED DESCRIPTION:
Obesity is a public health problem. Currently, the best treatment is surgery. However, 15% of patients after surgery have problems such as nausea, pain, vomiting, heartburn or regurgitation. To investigate these problems, an endoscopy is used. Yet, endoscopy has some disadvantages such as the need for intravenous sedation, need to take time off work, need for special endoscopy units and nurses and a delay in diagnosing because the endoscopy cannot be done at the time of the clinic visit. A new technology called clinic-based nasopharyngoendoscopy can potentially solve many of the problems with the current endoscopy. This study aims to determine that this new technology is just as effective in diagnosing problems as the current gold standard.

ELIGIBILITY:
Inclusion Criteria:

* Post-operative gastric bypass patients at St. Joseph's Healthcare Hamilton
* No previous nasal or pharyngeal surgery
* Foregut dyspeptic symptoms including: nausea, vomiting, regurgitation, epigastric pain, reflux and/or hematemesis
* Require endoscopy for investigation of foregut symptoms
* Able to provide consent

Exclusion Criteria:

* Patients who have not undergone gastric bypass surgery
* Inability to give consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-05; Primary Completion 2013-05 (Estimated); Study Completion 2013-05 (Estimated)

PRIMARY OUTCOMES:
Sensitivity, specificity, and positive and negative predictive values of in-office transnasal esophagoscopy in evaluating symptomatic, post-operative bariatric surgery patients. | Approximately 8 weeks
  The patients will receive transnasal esophagoscopy, then standard endoscopy approximately 2 weeks later. Patients will return to the bariatric clinic 2-4 weeks after standard endoscopy to review the results of both procedures and discuss possible treatment. Patients will not be required to undergo any further study-related follow-up or complete any questionnaires.

SECONDARY OUTCOMES:
Complications of standard and in-office transnasal esophagoscopy | approximately 8 weeks
  The patients will receive transnasal esophagoscopy, then standard endoscopy approximately 2 weeks later. Patients will return to the bariatric clinic 2-4 weeks after standard endoscopy to review the results of both procedures and discuss possible treatment. Patients will not be required to undergo any further study-related follow-up or complete any questionnaires.
Differences in in-hospital resource use between standard endoscopy and office-based transnasal nasopharyngoendoscopy | Approximately 8 weeks
  The patients will receive transnasal esophagoscopy, then standard endoscopy approximately 2 weeks later. Patients will return to the bariatric clinic 2-4 weeks after standard endoscopy to review the results of both procedures and discuss possible treatment. Patients will not be required to undergo any further study-related follow-up or complete any questionnaires.
How well patients tolerate in-office transnasal esophagoscopy | Immediately following transnasal esophagoscopy
  The patients will receive transnasal esophagoscopy, then standard endoscopy approximately 2 weeks later. Patients will return to the bariatric clinic 2-4 weeks after standard endoscopy to review the results of both procedures and discuss possible treatment. Patients will not be required to undergo any further study-related follow-up or complete any questionnaires.

CONTACTS AND LOCATIONS:
Overall Officials: Dennis Hong, MD, Principal Investigator — McMaster University
Locations (1):
- St. Joseph's Healthcare Hamilton, Hamilton, Ontario, Canada